CLINICAL TRIAL: NCT05599152
Title: A Study of Clinical Outcomes in Patients With Myocardial Infarction Who Maintained Novel Antiplatelet Agents for 1 Year and Patients Who Switched to Clopidogrel Early
Brief Title: Comparison of Myocardial Infarction Patients Who Were Prescribed a Novel Antiplatelet Agent or Clopidogrel
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chan Joon Kim (Other)
Collaborators: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor-Investigator, Chan Joon Kim, professor, Uijeongbu St. Mary Hospital
Organization: Uijeongbu St. Mary Hospital (Other)
Other Study IDs: CKD-HIRA-Data-Review
Record Dates: First submitted 2022-10-25; First posted 2022-10-31 (Actual); Last update posted 2022-10-31 (Actual); Status verified 2022-10

CONDITIONS: Myocardial Infarction
Keywords: clopidogrel; novel antiplatelet agent
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ticagrelor/prasugrel Group: Patients with acute myocardial infarction who underwent percutaneous coronary intervention and maintained aspirin and ticagrelor/prasugrel as standard therapy.
- clopidogrel Group: In patients with acute myocardial infarction who underwent percutaneous coronary intervention, discontinued ticagrelor/prasugrel and switched to clopidogrel

SUMMARY:
Myocardial infarction is defined according to icd-10 using the data base of South korea National Health Insurance Corporation, where personal identification information has already been removed, and detailed results are derived for each drug category.

DETAILED DESCRIPTION:
The purpose of this study is to compare the prognosis of patients with clopidogrel after early discontinuation of ticagrelor/prasugrel with patients who maintained aspirin and ticagrelor/prasugrel as standard therapy in patients with acute myocardial infarction who underwent percutaneous coronary intervention.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have a diagnosis code for acute myocardial infarction indicated in the National Health Insurance data and data for drugs that have used ticagrelor/prasugrel for 30-90 days when hospitalized for the relevant disease.
* Patients who switched to clopidogrel after 30-90 days.
* Patients with a diagnosis code for Venus myocardial infarction and a prescription code for percutaneous cardiovascular intervention in the National Health Insurance data.
* Adults 18 years of age or older

Exclusion Criteria:

* A person who has data for requesting blood transfusion during the period of hospitalization in the National Health Insurance data
* Those who have data for oral anticoagulants (warfarin, Coumadin, apixaban, edoxaban, dabigatran, rivaroxaban) in the National Health Insurance data
* Those who have a diagnosis code for malignant tumor in the National Health Insurance data
* Those who have end-stage renal failure code in the National Health Insurance data or those who have data for hemo/peritoneal dialysis
* A person who has a request for blood transfusion during the period of using Ticagrelor/prasugrel

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Prognostic data of patients who maintained aspirin and ticagreolor/prasugrel as standard therapy in patients with acute myocardial infarction who underwent percutaneous coronary intervention, and patients with clopidogrel after early discontinuation of ticagrerol/prasugrel
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2020-05-21 (Actual); Primary Completion 2022-11 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Composite of all-cause death, recurrent myocardial infarction, stroke, (ischemic and hemorrhagic ) and bleeding within one year. | Percutaneous coronary intervention after 1 Year
  compared patients who maintained ticagrelor/Prasugrel with those who switched from ticagrelor/prasugrel to clopidogrel.
  * All cause death
  * Myocardial infarction
  * Stroke
  * Bleeding
  Categorical data is indicated by number (%) and analyzed by X2 statistics. Continuous variables are expressed as mean standard deviation (±SD) , and in the case of skewed distribution, comparison is made by Mann-Whitney test or Student t test. To balance differences in baseline characteristics, stabilized inverse probability of treatment weighting (sIPTW) is used. For further analysis, consider propensity score matching (PSM) with nearest neighbor method and standardized mortality ratio weighting (SMRW) estimation.
  Propensity score uses a generalized additive logistic model and considers demographic data (age, gender, hypertension, diabetes mellitus, heart failure hemodialysis).

CONTACTS AND LOCATIONS:
Overall Officials: Chan Joon Kim, Principal Investigator — The Catholic University of Korea, Uijeongbu ST. Mary's Hospital
Locations (1):
- The Catholic University of Korea, Uijeongbu ST. Mary's Hospital, Uijeongbu-si, South Korea